CLINICAL TRIAL: NCT05808075
Title: Clinical Performance of Nano Fiber Reinforced Resin Composite Versus Conventional Nano Hybrid Resin Composite in Restoration of Compound Proximal Carious Lesions in Premolar Teeth: Two Years Randomized Clinical Trial
Brief Title: Clinical Performance of Nano Fiber Reinforced Versus Conventional Nano Hybrid Composite in Restoring Premolars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Raafat Abd-ElMoneim Hafez Khalid, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27722
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Clinical Performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NovaProTM Fill Universal Dental Composite (Experimental): NovaProTM Fill Universal Dental Composite will be selected , the tooth will be selectively etched with Phosphoric acid gel (37%) to enamel for 30 seconds .The etchant will be removed and the cavity will be rinsed with water spray for 30 seconds and air dried. A uniform thin layer of the adhesive will be applied on all the prepared surfaces then will be dispersed with a stream of air and then light cured. The restorative material will be applied using an incremental filling technique starting at the gingival wall. The restoration will be cured in 2 mm increments for 20 s. The proximal surfaces will be contoured with finishing strips following manufacturer's instructions. The occlusion will be checked with a thin articulating paper and will be adjusted by removing material with a fine diamond or stone. Finishing will be accomplished by finishing diamond stones then polished using rubber points
  Interventions: Other: NovaProTM Fill Universal Dental Composite
- Tetric N-Ceram Nano-hybrid Dental Composite (Active Comparator): The tooth will be selectively etched with N-Etch (IvoclarVivadent, Schaan, Liechtenstein) Phosphoric acid gel (37%) to enamel for 30 seconds. The etchant will be removed and the cavity will be rinsed with water spray for 30 seconds and dried with air syringe. A Uniform thin layer of the adhesive will be applied on all the prepared surface then dispersed with a stream of air and then light cured (Woodpecker Light Cure LED ,China).The restorative material Tetric N-Ceram Nano-hybrid will be applied using an incremental filling technique starting at the gingival wall. Each increment will be polymerized for 20 seconds., Occlusal adjustments will be made using articulating paper. Finishing will be accomplished by finishing diamond then polished using rubber points
  Interventions: Other: NovaProTM Fill Universal Dental Composite

INTERVENTIONS:
Other: NovaProTM Fill Universal Dental Composite — NovaProTM Fill Universal ,Nanova product

SUMMARY:
In patients that need composite restorations in a compound proximal carious lesions in premolars, will the clinical performance of nano fiber reinforced resin composite restorations have similar results compared to those restored with conventional nano hybrid resin composite over two years follow up period?

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University outpatient clinic. The operator in charge will be DR. The patients in this study will be selected according to different exclusion and inclusion criteria.

Teeth that meet the inclusion criteria will be selected (n=26) and divided into two groups (n=13).

Group (1): NovaProTM Fill Universal Composite (Nanova Columbia.MO. USA).Group (2): Tetric N-Ceram Nano-hybrid (IvoclarVivadent, Schaan, Liechtenstein). Teeth will be cleaned to remove surface stains. Compound proximal cavities will be prepared with rounded internal angles and with non beveled margins. The carious tissues will be removed using diamond burs of the suitable size at high speed under profuse water cooling system. After the cavity preparation and the appropriate shade of resin material selected, all restorations will be performed using a pre-curved metallic sectional matrix associated with a separating ring and a proper sized wooden wedge to establish the anatomical shape and proximal contacts of the teeth. All the restorative materials will be applied according to the manufacturer instructions (n=13)

All participants will be instructed to follow oral hygiene measures (brush the teeth twice a day, floss once a day) to avoid plaque and bacterial accumulation which may negatively affect the performance.

The restorations will be evaluated at baseline (after placement of restoration), after 6, 12, 18 & 24 months, using Modified United States Public Health Service criteria (USPHS) for the following characteristics: Anatomic Form (Wear), Marginal integrity, Surface roughness, Marginal discoloration, Color match, Recurrent caries, Post-operative sensitivity. The resin composite restorations will be evaluated with the aid of a dental explorer and an intraoral mirror and visual inspection. The restorations will be scored as follows: Alfa represents the ideal clinical situation, Bravo will be clinically acceptable and Charlie represents a clinically unacceptable situation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 18 to 55 years
* Male or Female patients
* Patients with good oral hygiene
* Patients with good recall availability

Exclusion Criteria:

* Patient who are allergic to products' ingredients used in the study
* Patients with poor oral hygiene
* Patients with history of bruxism and parafunctional habits
* Patients with high caries index or high plaque index.
* Pregnant or lactating women.
* History of severe medical complications such as xerostomia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Anatomic Form | 2 years
  Modified USPHS criteria United States Public Health Service
  USPHS criteria United States Public Health Service

SECONDARY OUTCOMES:
Mechanical, Esthetic and Biological properties | 2 years
  Modified USPHS criteria United States Public Health Service

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2025